CLINICAL TRIAL: NCT05467527
Title: Effectiveness of Prosocial-orientated Acceptance and Commitment Training (PACT) Programme for Parents of Children With Special Health Care Needs in Response to Outbreaks of Novel Infectious Disease: A Randomised Controlled Trial
Brief Title: PACT Programme for Parents of Children With SHCN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hong Kong Children's Hospital (Other); Hong Kong Young Women's Christian Association (Other)
Responsible Party: Principal Investigator, Yuen Yu CHONG, Assistant Professor, The Nethersole School of Nursing, CUHK, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2191269
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Urologic Diseases; Gastrointestinal Diseases; Vascular Diseases; Cleft Lip and Palate; Neurodevelopmental Disorders; Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorder; Developmental Delay
Keywords: Acceptance and Commitment Therapy; Randomised Controlled Trial; Special health care needs; novel infectious disease; prosociality
MeSH Terms: conditions — Urologic Diseases; Gastrointestinal Diseases; Vascular Diseases; Cleft Lip; Neurodevelopmental Disorders; Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder; Learning Disabilities

STUDY DESIGN:
Intervention Model Description: Parallel Assignment; repeated-measures 2-arm randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomisation procedure will be carried by a clerical staff who has no involvements in this project. For parents, all participants will use the same mobile app tentatively branded as "Calm Parents" but receive different assigned contents of the app.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACT Group (Experimental): A combination of 6 online modules and 4 group-based video conferencing sessions of Prosocial-orientated Acceptance and Commitment Training plus positive parenting advice via a mobile app across 12 weeks
  Interventions: Behavioral: Prosocial-orientated Acceptance and Commitment Training plus positive parenting advice
- Control Group (Placebo Comparator): A combination of 6 online modules and 4 group-based video conferencing sessions of daily parenting challenges in caring for a child with SHCN plus positive parenting advice via a mobile app across 12 weeks
  Interventions: Behavioral: Positive parenting advice

INTERVENTIONS:
Behavioral: Prosocial-orientated Acceptance and Commitment Training plus positive parenting advice — The PACT group will receive a combination of 6 online modules and 4 group-based video conferencing sessions of Prosocial-orientated Acceptance and Commitment Training plus positive parenting advice via a mobile app across 12 weeks. The modules will cover real-life scenarios of daily parenting challenges in caring for a child with SHCN, followed by age-appropriate positive parenting advice based on the Centers for Disease Control and Prevention guidelines. After going through the scenarios, parents will be audio/visually guided to participate in ACT activities, including mindfulness exercises, ACT metaphors and experiential exercises, which will be used to increase psychological flexibility.
  Arms: PACT Group
Behavioral: Positive parenting advice — The Control Group will receive a total of 6 online modules and 4 group-based video conferencing sessions in a closed group of 6-8, 60 minutes per session guided by a trained facilitator via the mobile app across 12 weeks. The online modules will provide identical contents to those in the PACT group, but no guided ACT metaphors or experiential exercises. The interaction sessions serve to review and discuss the contents of online modules, but without the contents related to ACT/prosociality.
  Arms: Control Group

SUMMARY:
This randomised controlled trial aims to determine the efficacy of a 12-week, smartphone-based Prosocial-orientated Acceptance and Commitment Training (PACT) programme plus age-appropriate positive parenting advice on the psychological flexibility, prosociality, parenting competence and family functioning with parents of children with special health care needs as well as the mental well-being of parent-child dyads over 12 months follow-up.

DETAILED DESCRIPTION:
Background: The caregiving burden experienced by parents of children with special health care needs (SHCN) is known to be significant, and its impact tends to be exacerbated when an outbreak of a novel infectious disease occurs. As shown in this coronavirus (COVID-19) pandemic, with the prolonged disruptions of individualised rehabilitation/supporting services which cannot be substituted by digital/remoted format and the unprecedented economic hardship, many parents of children with SHCN are under psychological distress, affecting parenting behaviours and child well-being. Existing interventions in literature only serve for suspected/infected cases/healthcare workers. Many interventions were developed without a conceptual understanding of what/how the proposed active/therapeutic ingredient(s)/process(es) could lead to desired outcomes. This study informs the development of a conceptual model, showing that two psychological constructs, namely psychological flexibility (a therapeutic process measured in Acceptance and Commitment Therapy) and prosociality (an attitude and/or behaviour that orient(s) toward the welfare of others and society) played significant roles in mitigating the adverse impact of COVID-19 on parental mental health.

Objectives: To determine the efficacy of a 12-week, smartphone-based Prosocial-orientated Acceptance and Commitment Training (PACT) programme plus age-appropriate positive parenting advice on the psychological flexibility, prosociality, parenting competence of parents and family functioning parents of children with SHCN as well as the mental well-being of parent-child dyads over 12 months follow-up.

Hypotheses to be tested: When compared to the Control Group, the participation in the PACT programme could improve parental mental well-being, child mental well-being, parental psychological flexibility and parental prosociality, parenting competence and family functioning at immediate, 3-, 6- and 12 months after the completion of the programme.

Design and subjects: A randomised controlled trial with a blinded, two-arm, repeated-measures design; 196 Cantonese-speaking parents/caregivers of children with special health care needs.

Study Instruments: Validated questionnaires.

Intervention: A 12-week, smartphone-based Prosocial-orientated Acceptance and Commitment Training (PACT) programme plus age-appropriate positive parenting advice.

Primary outcome measure: Parental mental well-being and child mental well-being.

Data analysis: Generalised estimating equation specifying an identity link function and a normal distribution will be employed to examine its change across two groups and all assessment time-points, followed by posthoc comparisons.

Expected results: To increase the mental well-being of parents and their children with special health needs. In addition, parenting competence and family functioning will also be improved.

ELIGIBILITY:
Inclusion Criteria:

* Cantonese-speaking Hong Kong residents
* Living together with the child who is at preschool/school-age (3-8 years old)
* Caregivers who adopted the responsibility of taking care of the child,
* has daily access to their iPhone and Android smartphones.

In addition, potential eligible parents who respond "yes" to any of the five validated screening questions in the Children with Special Health Care Needs (SHCN) Screener (see https://www.childhealthdata.org/docs/cshcn/technical-summary-of-cshcn-screener.pdf) will then be asked the associated follow-up questions to determine whether the child possesses physical, neurodevelopmental/emotional problem(s) that has lasted for at least 12 months. Only children with a positive response(s) to ≥ 1 item in each of the associated follow-up questions will be classified as children with SHCN.

Exclusion Criteria:

* Parents who have diagnoses of severe mental illness or developmental disabilities, such as intellectual disabilities

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Parental mental well-being | Change from baseline assessment to immediate, 3, 6 and 12 months post-intervention
  The 14-item Mental Health Continuum Short Form for Adults (MHC-SF) will be used to assess the emotional, social and psychological well-being of parents. MHC-SF can be scored between 0 and 5 (6 points Likert scale), which means that the total score on the scale can range from 0 to 70 points. Higher scores indicate a higher level of emotional wellbeing. scaleThe MHC-SF subscales possessed good convergent validity and internal consistencies in Western populations (Lamers et al., 2011).
Child mental well-being | Change from baseline assessment to immediate, 3, 6 and 12 months post-intervention
  The 25-item Strengths and Difficulties Questionnaire (SDQ, 25 items, 3-point Likert scale) will be adopted to evaluate the psychological adjustment of children with SHCN, in terms of conduct problems, hyperactivity, emotional symptoms, peer problems and prosocial behaviours. A total difficulties score can be generated by summing scores from all the scales except the prosocial scale. The resultant score ranges from 0 to 40. The SDQ is one of the most commonly used proxy reports from parents to assess the psychopathology of their children aged 3-16 years (Lai et al., 2010).

SECONDARY OUTCOMES:
Parental psychological flexibility | Change from baseline assessment to immediate, 3, 6 and 12 months post-intervention
  The 6-item PsyFlex (5-point Likert Scale) will assess all six therapeutic processes in Acceptance and Commitment Therapy (ACT). Each item refers to one of the core skills that ACT focuses on when developing psychological flexibility and well-being. The score is then interpreted such that higher scores represent higher psychological flexibility. (Hayes et al., 2011).
Parental prosociality | Change from baseline assessment to immediate, 3, 6 and 12 months post-intervention
  The 16-item Prosocialness Scale for Adults assesses 4 types of prosocial behaviours, including sharing, helping, taking care of, and feeling empathic with others from 1 (never/almost never) to 5 (almost always/always true) and summing all responses and finding the mean to get a total score (Caprara et al., 2005).
Parenting competence | Change from baseline assessment to immediate, 3, 6 and 12 months post-intervention
  The 17-item Chinese Version of the Parenting Sense of Competency Scale (C-PSOC; Ngai, Chan,& Holroyd E, 2007) will be used to assess parents' perceptions of their abilities to manage parenting needs. The PSOC comprises two subscales - the Efficacy subscale and the Satisfaction subscale. The Efficacy subscale contains eight items measuring parents' perception of competence in the parenting role. Differently, the Satisfaction subscale contains nine items evaluating the satisfaction and comfort of parents with the parenting role. Each item is scored using a 6-point Likert scale, ranging from 1 (strongly disagree) to 6 (strongly agree). The total score ranges from 17 to 102, while subscale scores range for the Efficacy and Satisfaction subscales are 17 to 48 and 17 to 54, respectively. The higher the score, the higher sense of competence and satisfaction in parenting. The PSOC had adequate internal consistencies (α=.77-.85) and test-retest reliabilities (r=.87) among Hong Kong parents.
Family functioning | Change from baseline assessment to immediate, 3, 6 and 12 months post-intervention
  The 36-item Chinese version of the Pediatric Quality of Life Inventory Family Impact Module (PedsQL FIM; Chen et al., 2011) will be adopted to assess the impact of pediatric asthma comorbid with ADHD on parent health-related quality of life and the family functioning. The PedsQL FIM consists of 8 subscales: Physical Functioning (6 items), Emotional Functioning (5 items), Social Functioning (4 items), Cognitive Functioning (5 items), Communication (3 items), Worry (5 items), Daily Activities (3 items) and Family Relationships (5 items). The former six subscales measure parents' overall functioning, while the latter two subscales measure parent-reported family functioning. Each item has five Likert response options, which are 0 (never a problem) to 4 (almost always a problem). Items are then linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0) and averaged by the number of items, so that higher scores indicate better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yuen Yu Chong, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Department of Surgery, Hong Kong Children's Hospital, Ngau Tau Kok, Kowloon
  - Hong Kong Young Women's Christian Association, Kowloon